CLINICAL TRIAL: NCT01286922
Title: The Insulin Sensitivity Using Aerobic Interval Conditioning
Acronym: ISAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 29018; R56DK081807 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Pre-diabetes
Keywords: diabetes; exercise; insulin resistance; interval training; physical activity
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus; Motor Activity; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interval Training (Experimental): The target intensity for the INT group is 2 min at about 95% of baseline VO2max followed by 2 min of recovery at 40-50% of VO2max. Regardless of the training method each participant will be "locked" into a weekly energy expenditure of 12 kilocalories per kilogram of body weight per week (KKW).
  Interventions: Other: Behavioral: exercise
- Aerobic Conditioning (Placebo Comparator): During the first AER training condition, we will train all participants at an energy expenditure of 12 kcal/kg/wk (KKW). The target exercise intensity for the AER group will be 50%-70% of baseline V02max.
  Interventions: Other: Behavioral: exercise

INTERVENTIONS:
Other: Behavioral: exercise — Specific Aim: We will identify, recruit, assess, and randomly assign 42 sedentary, overweight-obese individuals who are at risk for pre-diabetes to an AER or INT training group in order to test the hypothesis:
  • Individuals randomized to INT will have greater improvements in insulin sensitivity than individuals assigned to traditional AER.
  Secondary Aim: We will measure maximal cardiorespiratory fitness (VO2max/peak) in order to test the hypothesis:
  • Individuals randomized to the INT group will have a greater improvement in VO2max/peak than individuals in traditional AER group.

SUMMARY:
The Insulin Sensitivity using Aerobic Interval Conditioning (ISAIC) trial will compare traditional aerobic training (AER) to interval training (INT) in sedentary, overweight/obese men at risk for pre-diabetes. The investigators will randomly assign 42 individuals to 3 months of monitored exercise using a randomly assisgned design where participants will exercise under either AER or INT training conditions. The AER training condition will be consistent with "standard-of-care" recommendations. Exercise training will entail one 3-month blocks of either AER or INT. Training will consist of 1) a 1-month ramp up period, 2) 1-month of traditional aerobic training and 3) 1-month of either continued AER or INT.

DETAILED DESCRIPTION:
It is currently estimated that type II diabetes (T2D) affects 5-8% of adults. Also recognized is a transitional group of individuals whose control of blood glucose is abnormal, but not yet considered diabetic. These individuals are classified as having pre-diabetes, which is defined as having impaired fasting glucose (IFG;fasting glucose 100-125 mg/dl), impaired glucose tolerance (IGT; post 2-h glucose load; 140-199 mg/dl) or both. This population represents a significant segment of the population as it is estimated that approximately 23% of Americans have pre-diabetes (IGT or IFG). Two unifying features associated with these metabolic impairments is a strong link to obesity and physical inactivity. Regular exercise positively influences IFG/IGT and obesity, and represents an important therapy for preventing the progression to T2D by enhancing several mechanisms of action including improved: glucose metabolism, muscle respiratory capacity, mitochondrial respiratory chain activity and ß-oxidation. Importantly, the dose of physical activity required to promote metabolic benefits appears to be obtainable for most individuals with as little as ~1000 kcal/w of aerobic activity.

While most exercise policy statement guidelines recommend that exercise be performed within an intensity ranging of 40-85% V02max, newer guidelines, such as the recently updated Physical Activity and Public Health Recommendations recognize that few studies have examined the effects of intensity, duration, or frequency of physical activity independent of their contribution to the total amount of physical activity. Accordingly, this writing group specifically recommended that, "based on recent data, there is some indication that vigorous-intensity activities may have greater benefit for reducing cardiovascular disease and premature mortality than moderate-intensity physical activity .... that much more work is needed is this area."

ELIGIBILITY:
Inclusion Criteria:

* Age 30 to 60 years, inclusive
* BMI greater than or equal to 25 - less than or equal to 35 kg/m2
* Waist circumference >38"; Waist-to-Hip Ratio >0.95 Sedentary Lifestvle
* Not physically active greater than or equal to 3 days/week-l for 20 min each time for the previous 6 months,
* Not participating in regular resistance exercise

Exclusion Criteria:

* Resting blood pressure greater than or equal to 160/100 mm Hg
* Triglycerides greater than or equal to 500 mg/dL
* Factors that may limit adherence to intervention or affect conduct of the trial such as lack of time, amount of travel, and/or work or family stressors
* Unable or willing to communicate with staff, to provide written informed consent, or accept the randomized assignment
* Failure to complete behavioral run-in and baseline testing
* Hospitalization for depression in the last 6 months
* Not physically capable of performing the exercise required of the study protocols
* Consuming >14 alcoholic beverages per week
* Plans to be away >4 weeks in the next 6 months
* Lack of support from primary health care provider or family members
* Signficant weight loss in the past year (>20 kg) or current use of weight loss medications
* Current diagnsis of schizophrenia, or other psychotic disorders, or bipolar disorder
* Another member of household is a participant or staff member of the study.
* History of bariatric surgery within last 3 years,
* Other temporary intervening event, such as sick spouse, bereavement, or recent move.
* Other medical, psychiatric, or behavioral limitations that in the view of the principal investigator may interfere with study participation or the ability to follow the intervention protocol.
* Underlying diseases or conditions likely to limit lifespan and/or affect the safety of the intervention
* Cancers requiring treatment in the past 5 years, unless prognosis is excellent.
* Self-report HIV or tuberculosis.
* History or evidence of serious arrhythmias, cardiomyopathy, congestive heart failure, aortic aneurysm, or heart transplantation.
* Renal disease: currently receiving dialysis.
* Type I diabetes mellitus
* Type 2 diabetes mellitus, defined as:

Fasting plasma glucose levels greater than or equal to 26 mg/dL 2-hour postprandial Oral Glucose Tolerance Test results greater than or equal to 200 mg/dL

* Any other medical condition or disease that is life threatening or that can interfere with or be aggravated by exercise.
* Chronic obstructive lung disease, peripheral vascular disease or angina that limits ability to follow exercise protocol.
* Advanced neuropathy or retinopathy.
* Smoker or have used nicotine/tobacco products within the last 12 months.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 3 months
  Individulas randomized to INT will have greater improvements in insulin sensitivity than individuals assigned to traditional AER.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | 3 months
  Individuals randomized to the INT group will have a greater improvement in VO2max/peak than individuals in traditional AER group.

CONTACTS AND LOCATIONS:
Overall Officials: Conrad P. Earnest, PhD, Principal Investigator — Pennington Biomedical Research Center; Timothy S. Church, MD, MPH, PhD, Study Director — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Harris MI, Flegal KM, Cowie CC, Eberhardt MS, Goldstein DE, Little RR, Wiedmeyer HM, Byrd-Holt DD. Prevalence of diabetes, impaired fasting glucose, and impaired glucose tolerance in U.S. adults. The Third National Health and Nutrition Examination Survey, 1988-1994. Diabetes Care. 1998 Apr;21(4):518-24. doi: 10.2337/diacare.21.4.518. PMID 9571335
- [Background] Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Report of the expert committee on the diagnosis and classification of diabetes mellitus. Diabetes Care. 2003 Jan;26 Suppl 1:S5-20. doi: 10.2337/diacare.26.2007.s5. No abstract available. PMID 12502614
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2007 Jan;30 Suppl 1:S42-7. doi: 10.2337/dc07-S042. No abstract available. PMID 17192378
- [Background] Benjamin SM, Valdez R, Geiss LS, Rolka DB, Narayan KM. Estimated number of adults with prediabetes in the US in 2000: opportunities for prevention. Diabetes Care. 2003 Mar;26(3):645-9. doi: 10.2337/diacare.26.3.645. PMID 12610015
- [Background] Zierath JR, Tsao TS, Stenbit AE, Ryder JW, Galuska D, Charron MJ. Restoration of hypoxia-stimulated glucose uptake in GLUT4-deficient muscles by muscle-specific GLUT4 transgenic complementation. J Biol Chem. 1998 Aug 14;273(33):20910-5. doi: 10.1074/jbc.273.33.20910. PMID 9694838
- [Background] Lund S, Holman GD, Schmitz O, Pedersen O. Contraction stimulates translocation of glucose transporter GLUT4 in skeletal muscle through a mechanism distinct from that of insulin. Proc Natl Acad Sci U S A. 1995 Jun 20;92(13):5817-21. doi: 10.1073/pnas.92.13.5817. PMID 7597034
- [Background] Hayashi T, Wojtaszewski JF, Goodyear LJ. Exercise regulation of glucose transport in skeletal muscle. Am J Physiol. 1997 Dec;273(6):E1039-51. doi: 10.1152/ajpendo.1997.273.6.E1039. PMID 9435517
- [Background] Turcotte LP, Richter EA, Kiens B. Increased plasma FFA uptake and oxidation during prolonged exercise in trained vs. untrained humans. Am J Physiol. 1992 Jun;262(6 Pt 1):E791-9. doi: 10.1152/ajpendo.1992.262.6.E791. PMID 1319676
- [Background] Kiens B, Essen-Gustavsson B, Christensen NJ, Saltin B. Skeletal muscle substrate utilization during submaximal exercise in man: effect of endurance training. J Physiol. 1993 Sep;469:459-78. doi: 10.1113/jphysiol.1993.sp019823. PMID 8271208
- [Background] Gregg EW, Gerzoff RB, Caspersen CJ, Williamson DF, Narayan KM. Relationship of walking to mortality among US adults with diabetes. Arch Intern Med. 2003 Jun 23;163(12):1440-7. doi: 10.1001/archinte.163.12.1440. PMID 12824093
- [Background] Fletcher GF, Blair SN, Blumenthal J, Caspersen C, Chaitman B, Epstein S, Falls H, Froelicher ES, Froelicher VF, Pina IL. Statement on exercise. Benefits and recommendations for physical activity programs for all Americans. A statement for health professionals by the Committee on Exercise and Cardiac Rehabilitation of the Council on Clinical Cardiology, American Heart association. Circulation. 1992 Jul;86(1):340-4. doi: 10.1161/01.cir.86.1.340. No abstract available. PMID 1617788
- [Background] Physical activity and cardiovascular health. NIH Consensus Development Panel on Physical Activity and Cardiovascular Health. JAMA. 1996 Jul 17;276(3):241-6. PMID 8667571
- [Background] American College of Sports Medicine Position Stand. The recommended quantity and quality of exercise for developing and maintaining cardiorespiratory and muscular fitness, and flexibility in healthy adults. Med Sci Sports Exerc. 1998 Jun;30(6):975-91. doi: 10.1097/00005768-199806000-00032. PMID 9624661
- [Background] Albright A, Franz M, Hornsby G, Kriska A, Marrero D, Ullrich I, Verity LS. American College of Sports Medicine position stand. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2000 Jul;32(7):1345-60. doi: 10.1097/00005768-200007000-00024. PMID 10912903
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Result] Earnest CP, Lupo M, Thibodaux J, Hollier C, Butitta B, Lejeune E, Johannsen NM, Gibala MJ, Church TS. Interval training in men at risk for insulin resistance. Int J Sports Med. 2013 Apr;34(4):355-63. doi: 10.1055/s-0032-1311594. Epub 2012 Nov 23. PMID 23180210